CLINICAL TRIAL: NCT01796457
Title: HBRN: Immune Regulation and Costimulation in Natural History and Therapeutic Outcome of Chronic Hepatitis B
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kyong-Mi Chang, Professor, Gastroenterology, University of Pennsylvania
Other Study IDs: DK082864 Immunology Treatment; U01DK082864 (NIH)
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Immunology; HBV; Immune tolerant; Immune active
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an ancillary to the NIDDK-sponsored treatment trials titled: Combination Therapy of Pegylated Interferon Alfa-2a and Tenofovir Versus Tenofovir Monotherapy in Chronic Hepatitis B (NCT01369212) and Combination Entecavir and Peginterferon Therapy in HBeAg-Positive Immune-Tolerant Adults With Chronic Hepatitis B (NCT01369199).

This study will examine the balance between immune regulatory and effector responses in hepatitis B-infected participants enrolled in the HBRN's clinical trials (NCT01369212 and NCT01369199) to define natural history and treatment outcome.

DETAILED DESCRIPTION:
Aim 1. Therapeutic HBV suppression will enhance antiviral immune effector responses and reduce immune inhibitory factors in participants with chronic hepatitis B. This study will also examine if antiviral therapy has a durable effect in host immune phenotype and define the immunological effect of interferon-alpha (IFNα) therapy in chronic HBV participants.

Aim 2. Antiviral immune effector and regulatory responses before, during and/or after therapy can predict long term therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent for participation in the ancillary study

Exclusion Criteria:

* Children under 18 years of age
* Pregnant women
* Participants with anemia (Hgb<10 or Hct<30)
* Participants with active medical conditions such as congestive heart failure or chronic lung disease requiring oxygen, active coronary artery disease with unstable angina, sepsis and renal failure
* Participants with significant medical conditions, autoimmune disease or immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from multi-site clinical centers in the United States and Canada including primary care hospitals and community centers that have enrolled into the HBRN clinical trials (NCT01369212 or NCT01369199).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Immune regulatory and effector responses relative to HBV DNA, ALT and clinical outcome | up to 192 weeks
  HBV-specific lymphoproliferative, IFN-gamma and IL10 responses, T cell activation and costimulatory markers ( PD1, CTLA4, CD28, CD127), FoxP3+ Treg frequency, and NK frequency and expression of activating/inhibitory receptors Dendritic cell frequency

CONTACTS AND LOCATIONS:
Overall Officials: Kyong-Mi Chang, MD, Principal Investigator — University of Pennsylvania
Locations (8):
- United States (7):
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Plymouth, Minnesota
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
- Toronto Western Hospital Liver Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIDDK repository related to the study — https://repository.niddk.nih.gov/studies/hbrn-immunology-treatment/